CLINICAL TRIAL: NCT01095692
Title: Evaluating the Necessity of TOT Implantation in Women With Pelvic Organ Prolapse and Occult Stress Urinary Incontinence
Acronym: ATHENA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P090304
Record Dates: First submitted 2010-03-29; First posted 2010-03-30 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Stress Urinary Incontinence; Pelvic Organ Prolapse
Keywords: Occult stress Incontinence,; Pelvic Organ Prolapse,; Prevention of stress urinary incontinence,; Postoperative incontinence,; Sub-urethral tape
MeSH Terms: conditions — Urinary Incontinence, Stress; Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- only surgery (Active Comparator)
  Interventions: Procedure: Pelvic Organ Prolapse intervention
- surgery + TOT (Experimental)
  Interventions: Procedure: Pelvic Organ Prolapse and Suburethral TOT implantation

INTERVENTIONS:
Procedure: Pelvic Organ Prolapse and Suburethral TOT implantation — Procedure/Surgery: Pelvic Organ Prolapse intervention and Suburethral TOT implantation
  Other Names: Laparoscopic sacrocolpopexy; Vaginal surgery for prolapse using autologous tissue; Vaginal surgery for prolapse using synthetic mesh
  Arms: surgery + TOT
Procedure: Pelvic Organ Prolapse intervention — Procedure/Surgery: Pelvic Organ Prolapse intervention
  Other Names: -Laparoscopic sacrocolpopexy; -Vaginal surgery for prolapse using autologous tissue; -Vaginal surgery for prolapse using synthetic mesh
  Arms: only surgery

SUMMARY:
Nowadays the clinical significance of an occult stress urinary incontinence and its optimal treatment is not known.Regarding treatment, there are 2 main approaches : either the systematic preventive treatment of the occult stress urinary incontinence by means of a tension free vaginal tape (TOT) together with the treatment of prolapse or the treatment of prolapse in the first place and treatment of stress incontinence in a second time when and if it appears.This study is expected to provide objective evidence concerning the efficacy and security of TOT implantation for the prevention treatment of occult stress urinary incontinence in women with pelvic organ prolapse and occult urinary incontinence.The perspective is to improve the management of these patients by providing evidence based recommendation for their treatment.

DETAILED DESCRIPTION:
The study population consists of women with pelvic organ prolapse and occult stress urinary incontinence. They are randomised within two groups : one group with pelvic organ prolapse surgery alone and one group with implantation of TOT together with prolapse surgery for prevention of stress urinary incontinence.TOT implantation is performed as described previously, while the pelvic organ prolapse surgery could either be of abdominal (open or laparoscopic) or vaginal approach. Eighty eight (88) patients will be enrolled at 3 sites centers.

This study is a prospective, multicenter, randomised, active-control arm trial. The study population consists of women with pelvic organ prolapse and occult stress urinary incontinence. They are randomised within two groups : one group with pelvic organ prolapse surgery alone and one group with implantation of TOT together with prolapse surgery for prevention of stress urinary incontinence.TOT implantation is performed as described previously, while the pelvic organ prolapse surgery could either be of abdominal (open or laparoscopic) or vaginal approach. Eighty eight (88) patients will be enrolled at 3 sites centers.

Visit I (J-2 months +/- 1 month) :

During this visit the following will be performed :

* Collection of general medical, obstetric and surgical history of the patients
* Collection of incontinence, prolapse and sexual history with the following questionnaires :

  * Standard Questionnaire
  * PFIQ-7 : Pelvic Floor Impact Questionnaire
  * PFDI-20 : Pelvic Floor Distress Inventory-short version Questionnaire
  * PISQ-12 : Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire
* Clinical examination that includes :

  * a stress test in lithotomy position before and after reduction of prolapse with bladder filled with 250 cc of water. The reduction of prolapse will be performed manually and using a vaginal speculum. The results after both types of reduction will be recorded separately
  * a Vaginal examination establishing the oestrogen status of patient's vagina and classification of prolapse using Baden Walker halfway method and modified ICS POP-Q system
  * Urodynamic test that includes Uroflowmetry as follows :
  * urethral pressure profile, maximum urethral closure pressure (MUCP) and Valsalva leak point pressure (VLPP) determination before and after reduction of prolapse manually
  * Filling cystometry without reduction of prolapse Post void residual volume of urine will be recorded
  * Explanation of the research protocol
  * Evaluation criteria for inclusion and exclusion
  * Information and signed informed consent of the patient
  * Randomization

Hospitalization (J0 at J 6days +/- 2 days) :

During the stay in the hospital the following will be recorded:

* Type and duration of each procedure
* Total number of days of hospitalization
* Immediate complications (e.g perioperative hemorrhage requiring transfusion or not, urine retention requiring catheterisation)
* Postvoid residual volume of urine for all the patients by bladder scan

Visit II (J 45 days +/- 15 days) :

During this visit the following will be performed :

* Objective and subjective evaluation of POP treatment and TOT placement
* Filling out questionnaires :

  * PFIQ-7 : Pelvic Floor Impact Questionnaire
  * PFDI-20 : Pelvic Floor Distress Inventory-short version Questionnaire
* Clinical examination including :

  * Stress test in lithotomy position as of visit I
  * Vaginal examination
  * In case of prolapse, the modified ICS POP-Q and Baden Walker halfway method for quantification

Visit III (J 6 months +/- 1 month) :

During this visit the following will be performed :

* Filling out questionnaires :

  * PFIQ-7 : Pelvic Floor Impact Questionnaire
  * PFDI-20 : Pelvic Floor Distress Inventory-short version Questionnaire
  * PISQ-12 : Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire
  * PGI-I : Patient Global Impression of Improvement
  * Degree of satisfaction by the operation (visual 0-10 scale)
* Clinical examination including :

  * Stress test in lithotomy position as of visit I
  * Vaginal examination
  * In case of prolapse, the modified ICS POP-Q and Baden Walker halfway method for quantification
* Uroflowmetry
* Short time pad test
* Full urodynamic test in case of incontinence or obstruction

ELIGIBILITY:
Inclusion Criteria:

* Female patients, at least 18 years of age
* Having a pelvic organ prolapse and occult stress urinary incontinence
* Patient non opposed to the exploitation of data in research
* Agree to comply with all protocol-specified procedures, including protocol mandated follow up visits

Exclusion Criteria:

* Symptoms of stress urinary incontinence preoperatively
* Patients not having social security
* Pregnancy or lactation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
To compare the postoperative prevalence of stress incontinence in patients with or without TOT implant during a pelvic organ prolapse surgery | 6 month

SECONDARY OUTCOMES:
To compare the severity of postoperative stress urinary incontinence between the two groups | 6 month
To compare the prevalence of new onset overactive bladder postoperatively between the two groups | 6 month
To compare the severity of new onset overactive bladder between the two groups | 6 month
To compare the prevalence of postoperative dyspareunia at 6 months between the two groups | 6 month
To compare the prevalence of postoperative urinary retention between the two groups | 6 month
To compare the severity of postoperative dyspareunia at 6 months between the two groups | 6 month
To compare the prevalence of dyschesia and constipation at 6 months between the two groups | 6 month
To compare pre- and postoperative urodynamic test of patients when they are incontinent at 6 months | 6 month
To compare the postoperative Patient Global Impression of Improvement and degree of satisfaction at 6 months between the 2 groups | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Ariane Cortesse, MD, Principal Investigator — Department of Urology, Saint Louis Hospital
Locations (1):
- Diaconesses Hospital, Paris, Île-de-France Region, France

REFERENCES:
- [Result] Cortesse A, Jacquetin B, Grise P, Le Normand L, Richard F, Haab F. Prospective multicenter clinical trial of Uretex Sup for surgical treatment of stress urinary incontinence. Int J Urol. 2007 Jul;14(7):611-5. doi: 10.1111/j.1442-2042.2007.01542.x. PMID 17645604
- [Derived] Yeung E, Baessler K, Christmann-Schmid C, Haya N, Chen Z, Wallace SA, Mowat A, Maher C. Transvaginal mesh or grafts or native tissue repair for vaginal prolapse. Cochrane Database Syst Rev. 2024 Mar 13;3(3):CD012079. doi: 10.1002/14651858.CD012079.pub2. PMID 38477494
- [Derived] Maher C, Yeung E, Haya N, Christmann-Schmid C, Mowat A, Chen Z, Baessler K. Surgery for women with apical vaginal prolapse. Cochrane Database Syst Rev. 2023 Jul 26;7(7):CD012376. doi: 10.1002/14651858.CD012376.pub2. PMID 37493538